CLINICAL TRIAL: NCT01114906
Title: Estimating the Use of Resources and the Costs of Treating Patients With Asthma in the Autonomous Community of Valencia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RES-DUM-2010/1
Record Dates: First submitted 2010-04-20; First posted 2010-05-03 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Asthma; Valencia Autonomous Region
Keywords: Asthma; Resource use
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study has been conceived in the context of Health Outcomes Research where the outcomes of health interventions in routine clinical practice constitute the main objective of the research process. In the case of asthma in Spain, the investigators do not clearly know the use of resources generated by the patient with asthma, its impact on the effectiveness of the current approach of asthmatic patients and the overall efficiency of health interventions on asthmatic patients. This observational, retrospective and multicenter study aims to estimate the use of health care resources in managing patients with asthma and to determine the management of the disease in the usual clinical practice in Valencia Autonomous Region. The data will be obtained at primary care level from the Electronic Health Record SIA+GAIA data base and at hospital level from allergologists and pneumologists clinical records. The investigators plan to introduce 289 ambulatory patients followed-up in Primary or Specialized Care Services, older than 15 years of age, diagnosed of asthma at least one year before the beginning of the study. The inclusion period will be of 3 months and the retrospective data of 12 previous months of follow-up will be collected.

The direct and indirect use of resources will be collected in order to estimate the management and use of health care resources in managing patients with asthma in the Autonomous region of Valencia as primary endpoint and also to estimate the mean cost of asthmatic patient healthcare; to determine the global effectiveness and the efficiency of the actual asthmatic patient healthcare and to model the health budget according to different objectives of effectiveness for the next five years.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients (Primary and Specialized Care)
* Patients with a diagnose of asthma in the Outpatients' Electronic Health Record [Historia Clínica Ambulatoria electrónica (SIA + GAIA) database

Exclusion Criteria:

* Patients who have participated in a clinical trial in the last 12 months.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ambulatory patients followed-up in Primary or Specialized Care Services (hospital)
Sampling Method: Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Direct and indirect Resource Use of Asthma patients in 12 months | Once the patient has been included data refered to the previous 12 month following-up period will be recorded. Thus, all data will be recorded at that time-period. Only one data recording will be done.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Research Site, Alcoy, Alicante
  - Research Site, Vila-real, Castellón
  - Research Site, Valencia, Valencia
  - Research Site, Xàtiva, Valencia